CLINICAL TRIAL: NCT04429867
Title: Hydroxychloroquine Use in Hospitalized Patients With COVID-19: Impact on Progression to Severe or Critical Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: WellStar Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1604885
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine (Experimental)
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine 400 mg PO BID x 2 doses, then 200 mg PO BID x 8 doses
  Arms: Hydroxychloroquine
Drug: Placebo — Placebo 400 mg PO BID x 2 doses, then 200 mg PO BID x 8 doses
  Arms: Placebo

SUMMARY:
The primary objective is to assess the impact of hydroxychloroquine in hospitalized patients with COVID-19 and risk factors for severe/critical disease.

DETAILED DESCRIPTION:
This study will utilize a randomized, placebo-controlled, double-blinded design. Patients admitted with confirmed COVID-19, and at least 1 of the following: requiring oxygen supplementation (≤4 liters of oxygen via nasal cannula or increase from baseline), bilateral infiltrates on CT/CXR, age >65, diabetes, hypertension, BMI > 35, chronic lung disease, cardiovascular disease, chronic kidney disease, cancer (hematologic malignancies, lung cancer, and metastatic disease), will be randomized in a 1:1 fashion to hydroxychloroquine 400 mg PO BID x 2 doses, then 200 mg PO BID x 8 doses or placebo at a matching schedule.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Wellstar Kennestone Hospital
* Age 18 years or older
* Laboratory-confirmed COVID-19
* At least 1 of the following:

  1. Requiring oxygen supplementation at ≤ 4 liters via nasal cannula or increase from baseline
  2. Bilateral infiltrates on CXR or CT of chest
  3. Age 65 or older
  4. Diabetes
  5. Hypertension
  6. BMI > 35
  7. Chronic lung disease
  8. Cardiovascular disease
  9. Chronic kidney disease
  10. Cancer (hematologic malignancies, lung cancer, and metastatic disease)

Exclusion Criteria:

* Unable to provide informed consent
* Unable to take oral medication
* Severe/critical COVID-19 disease at presentation

  1. Intensive care or intermediate care required at admission or within 48 hours
  2. Requiring oxygen supplementation via high flow nasal cannula, bipap, or non-rebreather mask at admission or within 48 hours
* Likelihood of survival <48 hours in the opinion of the primary physician or transitioned to comfort measures within 48 hours of admission
* Inability to take hydroxychloroquine due to allergy, QTc > 500 ms (male) or 520 ms (female) prior to initiation of hydroxychloroquine, pre-existing retinopathy, known G6PD deficiency, known porphyria, or significant drug- drug interactions
* Pregnant or breastfeeding
* Severe liver disease (Child-Pugh Class C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-12-07 (Estimated); Study Completion 2020-12-07 (Estimated)

PRIMARY OUTCOMES:
Impact of hydroxychloroquine in hospitalized patients with COVID-19 and risk factors for severe/critical disease. | 30 Days
  The impact will be evaluated by comparing rates of a composite primary outcome in patients randomized to hydroxychloroquine versus those randomized to placebo. The composite outcome includes progression to severe/critical disease or death (including withdrawal of care/hospice transfer). Progression to severe/critical disease is defined by requiring oxygen delivery via high flow nasal cannula, non-rebreather mask, bipap, or transfer to intensive care (ICU) or intermediate care units (IMCU) due to COVID-19-related complications.

SECONDARY OUTCOMES:
Hospital length of stay | 30 Days
30-Day Mortality | 30 Days
Resolution of Symptoms | 14 Days
  Resolution of symptoms will be assessed using standard medical interview procedures with the subject and review of the medical records.
Incidence of QTc >500ms after initiation of therapy | 30 Days
Incidence of discontinuation of therapy | 30 Days

CONTACTS AND LOCATIONS:
Locations (1):
- Wellstar Kennestone Hospital, Marietta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No